CLINICAL TRIAL: NCT00832572
Title: A Double-blind, Placebo-controlled, Cross-over Study of Ranolazine in Patients With Coronary Artery Disease for the Treatment of Painful Polyneuropathy
Brief Title: Study of Ranexa in Patients With Coronary Artery Disease and Painful Polyneuropathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT 3042
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease; Pain; Peripheral Nervous System Diseases; Polyneuropathy
Keywords: Coronary Artery Disease; Pain; Peripheral Neuropathy; Polyneuropathy
MeSH Terms: conditions — Coronary Artery Disease; Pain; Peripheral Nervous System Diseases; Polyneuropathies | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo-Ranolazine (Experimental): Participants were randomized to receive placebo to match ranolazine during Weeks 1 to 6, then ranolazine during Weeks 7 to 12.
  Interventions: Drug: Ranolazine; Drug: Placebo
- Ranolazine-Placebo (Experimental): Participants were randomized to receive ranolazine during Weeks 1 to 6, then placebo to match ranolazine during Weeks 7 to 12.
  Interventions: Drug: Ranolazine; Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine ER tablet administered orally for 6 weeks (500 mg twice a day for 3 weeks, followed by either 500 mg or 1000 mg twice a day for 3 weeks).
  Other Names: Ranexa
Drug: Placebo — Placebo to match ranolazine administered twice a day for 6 weeks

SUMMARY:
This study was to determine whether ranolazine was effective in the treatment of neuropathic pain in patients with coronary artery disease.

Eligibility required neurological examination by the study doctor and assessment of the patient's pain. Eligible participants were randomized to receive blinded study medication for a total of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years
* Coronary artery disease with a clinically diagnosed peripheral neuropathy
* Willing and able to provide signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Willing and able to comply with the requirements of the protocol and follow directions from the clinic staff

Exclusion Criteria:

* History of allergy or intolerance to ranolazine
* Any condition or concomitant medication that would have precluded the safe use of ranolazine as outlined in the prescribing information sheet (see Appendix E)
* In the judgment of the investigator, any clinically-significant ongoing medical condition that might jeopardize the patient's safety or interfere with the absorption, distribution, metabolism or excretion of the study drug
* In the judgment of the investigator, clinically-significant abnormal physical findings during screening (excluding the patient's peripheral neuropathy condition)
* Use of any experimental or investigational drug or device within 30 days prior to screening
* Pregnant or breast feeding, or (if premenopausal), not practicing an acceptable method of birth control (as detailed in Inclusion Criterion 4)
* Had received prior treatment with, or investigational exposure to, ranolazine within 7 days prior to randomization
* Clinically significant hepatic impairment
* Had end-stage renal disease requiring dialysis
* Psychological or addictive disorders (not limited to, but including drug and/or alcohol dependency) that may have precluded patient consent or compliance, or that may have confounded study interpretation
* Positive pregnancy test at Baseline (pre-randomization, Day 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Walker, MD, Principal Investigator — Cardiovascular Institute of the South Clinical Research Corporation
Locations (1):
- Cardiovascular Institute of the South Clinical Research Corporation, Houma, Louisiana, United States

REFERENCES:
- See also: The Neuropathy Association, a public, non-profit organization providing information and support for patients with neuropathy — http://www.neuropathy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants were enrolled and treated.
Groups:
- Placebo/Ranolazine: Participants were randomized to receive placebo to match ranolazine during Weeks 1 to 6 (Period 1), then ranolazine (500 mg twice a day for 3 weeks, followed by either 500 mg or 1000 mg twice a day for 3 weeks) during Weeks 7 to 12 (Period 2).
- Ranolazine/Placebo: Participants were randomized to receive ranolazine (500 mg twice a day for 3 weeks, followed by either 500 mg or 1000 mg twice a day for 3 weeks) during Weeks 1 to 6 (Period 1), then placebo to match ranolazine during Weeks 7 to 12 (Period 2).
Period: Period 1
Arm/Group | Placebo/Ranolazine | Ranolazine/Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Placebo/Ranolazine | Ranolazine/Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Ranolazine | Ranolazine/Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Neuropathic Pain
Description: Reduction in patient-reported neuropathic pain (by 2 numeric levels as measured by the Numeric Pain Scale)
Time Frame: Baseline to Week 6
Population: Study was stopped and no analysis was performed on the primary outcome measure.
Arm/Group | Placebo/Ranolazine | Ranolazine/Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Assess Participant Quality of Life Utilizing the Short Form 36 Health Survey (SF-36v2) Questionnaire
Description: The participant quality of life assessed utilizing the SF-36v2 questionnaire
Time Frame: Baseline to Week 6
Population: Study was stopped and no analyses were performed on the secondary outcome measures.
Arm/Group | Placebo/Ranolazine | Ranolazine/Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Response to Thermal and Mechanical Stimuli
Description: The participant response to thermal and mechanical stimuli as measured by the Hargreaves and Von Frey tests
Time Frame: Baseline to Week 6
Population: Study was stopped and no analyses were performed on the secondary outcome measures.
Arm/Group | Placebo/Ranolazine | Ranolazine/Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Groups:
- Placebo/Ranolazine, Period 1: Adverse events for this reporting group are those occurring during Period 1 (participants were receiving placebo).
  Participants were randomized to receive placebo to match ranolazine during Weeks 1 to 6 (Period 1), then ranolazine (500 mg twice a day for 3 weeks, followed by either 500 mg or 1000 mg twice a day for 3 weeks) during Weeks 7 to 12 (Period 2).
- Placebo/Ranolazine, Period 2: Adverse events for this reporting group are those occurring during Period 2 (participants were receiving ranolazine).
  Participants were randomized to receive placebo to match ranolazine during Weeks 1 to 6 (Period 1), then ranolazine (500 mg twice a day for 3 weeks, followed by either 500 mg or 1000 mg twice a day for 3 weeks) during Weeks 7 to 12 (Period 2).
- Ranolazine/Placebo, Period 1: Adverse events for this reporting group are those occurring during Period 1 (participants were receiving ranolazine).
  Participants were randomized to receive ranolazine (500 mg twice a day for 3 weeks, followed by either 500 mg or 1000 mg twice a day for 3 weeks) during Weeks 1 to 6 (Period 1), then placebo to match ranolazine during Weeks 7 to 12 (Period 2).
- Ranolazine/Placebo, Period 2: Adverse events for this reporting group are those occurring during Period 2 (participants were receiving placebo).
  Participants were randomized to receive ranolazine (500 mg twice a day for 3 weeks, followed by either 500 mg or 1000 mg twice a day for 3 weeks) during Weeks 1 to 6 (Period 1), then placebo to match ranolazine during Weeks 7 to 12 (Period 2).
Arm/Group | Placebo/Ranolazine, Period 1 | Placebo/Ranolazine, Period 2 | Ranolazine/Placebo, Period 1 | Ranolazine/Placebo, Period 2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Ranolazine, Period 1 (N=3) | Placebo/Ranolazine, Period 2 (N=3) | Ranolazine/Placebo, Period 1 (N=2) | Ranolazine/Placebo, Period 2 (N=2)
Fever (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Sensitivity to light (eyes) (Nervous system disorders) | 0 | 0 | 0 | 1
Right leg muscle tendon pulled (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Stabbing pain to right leg calf (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Aching pain to right calf (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Expiratory wheezing (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was stopped after 5 participants were enrolled. No outcome measure analyses were performed. Adverse events were collected and reported to the study center's Institutional Review Board.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years